CLINICAL TRIAL: NCT04685096
Title: Efficacy Evaluation of the Anti-ageing Effect of a Cosmetic Active Versus Placebo
Brief Title: Anti-ageing Efficacy of a Cosmetic Formulation Containing NMN (2%) Versus Placebo
Status: Completed | Type: Observational
Sponsor: Seneque SA (Industry)
Collaborators: Eurofins (Industry); LGD (Industry)
Responsible Party: Sponsor
Other Study IDs: 19E4487
Record Dates: First submitted 2020-12-11; First posted 2020-12-28 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2020-12

CONDITIONS: Wrinkle; Fatigue; Puffiness Around the Eyes
Keywords: Skin aging
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asian skin: Twice-daily application for 55 Days
  Interventions: Other: Test product creme; Other: Reference creme
- African-American skin: Twice-daily application for 55 Days
  Interventions: Other: Test product creme; Other: Reference creme

INTERVENTIONS:
Other: Test product creme — twice daily application of creme containing 2% NMN
Other: Reference creme — twice daily application of reference creme

SUMMARY:
The study aims at evaluating skin wrinkling, puffiness and fatigue and dark circle appearance on asian and african-american healthy volunteer cohorts receiving a cosmetic formulation containing NMN (2%). The product will be evaluated after 28 and 56 days of twice-daily application in comparison with a reference cosmetic formulation using clinical scoring under dermatological control. Cosmetic acceptability and future use will also be subjectively evaluated by analysis of the subjects answers to an evaluation questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject
* Subject having given her free informed, written consent
* Subject willing to adhere to the protocol and study procedures
* Subject with normal frontal temperature lower than 37.5°c/100.4°F
* Subject has read and understood the information given by the investigator related to protection against Novel Coronavirus 19 and necessity to contact the investigator in case of any suspicion of COVID related manifestation (increase of frontal temperature, cough, sore muscles, weakness…) during the study

Exclusion Criteria:

* Pregnant or nursing woman or woman planning to get pregnant during the study
* Start, stop or change in hormonal treatment (including contraceptive pill) <1.5 months
* Cutaneous pathology on the study zone (face)
* Use of topical or systemic treatment during the previous weeks liable to interfere with the assessment of the cutaneous efficacy of the study product
* Subject having undergone a surgery under general anesthesia within the previous month
* Know allergy to certain cosmetic or dermato-pharmaceutic products
* Subject having done injections on face and/or a lifting
* Excessive exposure to sunlight or UV-rays within the month preceding the study

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type: Chinese and Afro-American subjects
  * In each group, 50% of the subjects will have normal skin, 50% will have mild dry skin (declarative)
  * 100% will have wrinkles or fine lines on the crow's feet
  * 50% will have dark circles (half of them in the Active group, half of them in the Placebo group)
  * 50% will have puffiness (half of them in the Active group, half of them in the Placebo)
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Wrinkles | Change from baseline (day 0) at days 28 and 56 of application
  clinical grading under dermatological control using 1) a 7 points Visual scale of Bazin from absence (0) to pronounced wrinkles (6) for the Asian panel and 2) a 5 points Visual scale of Bazin from absence (0) to pronounced wrinkles (4) for the Afro-American panel
Eye bags | Change from baseline (day 0) at days 28 and 56 of application
  clinical grading under dermatological control using 1) a 7 points Visual scale of Bazin from absence (0) to pronounced bags (6) for the Asian panel and 2) a 6 points Visual scale of Bazin from absence (0) to pronounced bags (5) for the Afro-American panel
Dark circles | Change from baseline (day 0) at days 28 and 56 of application
  clinical grading under dermatological control using 1) a 6 points Visual scale of Dermscan from absence (0) to important dark circles (6) for the Asian panel and 2) a 5 points Visual scale of Dermscan from absence (0) to important dark circles (4) for the Afro-American panel
Relaxed features | Change from baseline (day 0) at days 28 and 56 of application
  clinical grading under dermatological control using a 11 points Non structured scale from relaxed features (0) to looking tired (10) for both panels

SECONDARY OUTCOMES:
Subjective evaluation of the product agreeableness and its effects on skin texture, moisture, puffiness, brightness, youth, swelling, wrinkling, radiance and tone. | At day 28 of application
  Self-assessment questionnaire on a 5 points scale from "I disagree" (-2) to "I agree" (+2).
Subjective evaluation of the product agreeableness and its effects on skin texture, moisture, puffiness, brightness, youth, swelling, wrinkling, radiance and tone. | At day 56 of application
  Self-assessment questionnaire on a 5 points scale from "I disagree" (-2) to "I agree" (+2).

CONTACTS AND LOCATIONS:
Overall Officials: Corinne BENIER, Study Director — Dermscan
Locations (2):
- Eurofins CRL Cosmetics Inc, Piscataway, New Jersey, United States
- Eurofins China, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No